CLINICAL TRIAL: NCT02263456
Title: An Open Study to Compare the Pharmacokinetics and Safety of Replenine®-VF and Replenine® or Any Other High Purity Factor IX Concentrate, in Severe Haemophilia B Patients.
Brief Title: A Study to Compare the Pharmacokinetics and Safety of Replenine®-VF, Replenine® or Other Factor IX in Haemophilia B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: RP9VFPK
Record Dates: First submitted 2014-09-02; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-08

CONDITIONS: Haemophilia B
MeSH Terms: conditions — Hemophilia B

ARMS (2):
- Current Factor IX (Active Comparator)
  Interventions: Biological: Replenine®-VF (High Purity Factor IX)
- Replenine®-VF (Experimental)
  Interventions: Biological: Replenine®-VF (High Purity Factor IX)

INTERVENTIONS:
Biological: Replenine®-VF (High Purity Factor IX)

SUMMARY:
The purpose of this study is:

* to compare the pharmacokinetics of Replenine®-VF and Replenine® or any other high purity Factor IX concentrate, when given as a bolus dose of 75IU/kg.
* to compare the 1st and 2nd pharmacokinetic assessments on Replenine®-VF (conducted 3 months apart) and recovery if patients changes batches.
* to evaluate Replenine®-VF in terms of clinical tolerance and safety in patients with severe haemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 years or over
* At least 20 exposures suffering from severe Haemophilia B and without inhibitors to Factor IX and on Replenine® or any other high purity Factor IX product

Exclusion Criteria:

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-07; Primary Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration/time curve (AUC) for plasma Factor IX | Pre-dose, 10, 30 min, 1, 3, 6, 9, 12, 24, 30, 36, 50, 56 hr post-dose

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - The Royal Free Hospital, Pond Street, Hampstead, London
  - The North Hampshire Hospital, Aldermaston Road, Basingstoke
  - Addenbrooke's Hospital, Hills Road, Cambridge
  - University Hospital of Wales, Health Park, Cardiff
  - Kingston General Hospital, Beverly Road, Hull
  - Leicester Royal Infirmary, Infirmary Square, Leicester
  - Lincoln County Hospital, Greetwell Road, Lincoln

REFERENCES:
- See also: Related Info — http://www.bpl.co.uk